CLINICAL TRIAL: NCT03172338
Title: Smart - Systems Medicine of Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: German Heart Institute (Other)
Responsible Party: Sponsor
Other Study IDs: SMART
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The onset and course of heart failure (HF) is triggered by a complex regulatory network that includes stressors (pressure overload by individual anatomic hemodynamic settings), intrinsic (genes), environmental (regulating epigenetics), and modifying factors (such as hor-mones and the immune system). SMART aims to establish individualized strategies for the prevention and management of HF by early detection of the physiological, genomic, proteo-mic and hemodynamic mechanisms that lead from onecommon cause of ventricular dysfunction (pressure overload) to maladaptive remodelling and irreversible HF. To cope with the complexity of HF, SMART will interrelate models describing the interplay between ge-nome, proteome and cell function, regulating hormones, tissue composition and hemody-namic whole organ function up to a whole body description of a patient and patient cohorts. The ultimate goal is to demonstrate proof-of-concept tools for predicting disease evolution and efficacy of treatment in a given patient. To achieve this task SMART will apply

* A modelling framework that couples multi-scale mechanistic models with in-depth genome/proteome, cell physiology and whole organ (biomechanical and fluid dynamic) models
* Subsequently, investigate methods validity and relevance for "quantitative prediction" of treatment outcome in a clinical proof-of-concept trial (demonstrator) of patients with aortic valve desieases.

ELIGIBILITY:
Inclusion Criteria:

* Aortic Valve Stenosis

Exclusion Criteria:

* coronary heart disease

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinically relevant Aortic Valve Stenosis, who are scheduled for surgical Aortic Valve Replacement.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-06-02 (Actual); Primary Completion 2018-02-28 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
Hypertrophy | 3 months
  Muscle Mass and Fibrosis

CONTACTS AND LOCATIONS:
Locations (1):
- German Heart Center Berlin, Berlin, Germany

REFERENCES:
- [Derived] Berndt N, Eckstein J, Wallach I, Nordmeyer S, Kelm M, Kirchner M, Goubergrits L, Schafstedde M, Hennemuth A, Kraus M, Grune T, Mertins P, Kuehne T, Holzhutter HG. CARDIOKIN1: Computational Assessment of Myocardial Metabolic Capability in Healthy Controls and Patients With Valve Diseases. Circulation. 2021 Dec 14;144(24):1926-1939. doi: 10.1161/CIRCULATIONAHA.121.055646. Epub 2021 Nov 11. PMID 34762513
- [Derived] Nordmeyer S, Lee CB, Goubergrits L, Knosalla C, Berger F, Falk V, Ghorbani N, Hireche-Chikaoui H, Zhu M, Kelle S, Kuehne T, Kelm M. Circulatory efficiency in patients with severe aortic valve stenosis before and after aortic valve replacement. J Cardiovasc Magn Reson. 2021 Mar 1;23(1):15. doi: 10.1186/s12968-020-00686-0. PMID 33641670
- [Derived] Nordmeyer S, Hellmeier F, Yevtushenko P, Kelm M, Lee CB, Lehmann D, Kropf S, Berger F, Falk V, Knosalla C, Kuehne T, Goubergrits L. Abnormal aortic flow profiles persist after aortic valve replacement in the majority of patients with aortic valve disease: how model-based personalized therapy planning could improve results. A pilot study approach. Eur J Cardiothorac Surg. 2020 Jan 1;57(1):133-141. doi: 10.1093/ejcts/ezz149. PMID 31131388